CLINICAL TRIAL: NCT03136250
Title: Effects of Autogenic and Reciprocal Inhibition, Muscle Energy Techniques in the Management of Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUI/CTR/2017/1
Record Dates: First submitted 2017-04-10; First posted 2017-05-02 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2017-12

CONDITIONS: Neck Pain
Keywords: Muscle Energy Techniques; Autogenic Inhibition; Reciprocal Inhibition; Stretching; Range of Motion; Muscle Strength; VAS; Neck Disability Index; NDI
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: A randomized Controlled trial will be conducted in order to find and compare the effectiveness of conventional stretching and MET stretching (autogenic inhibition and reciprocal inhibition). One Control group (conventional group) and two Experimental groups (Experimental Group A - Autogenic Inhibition & Experimental Group B - Reciprocal Inhibition) will be formed. The participants will be recruited in the study if they meet the inclusion criteria using consecutive sampling from Fauji Foundation Hospital and randomized into the three respective groups. All the groups will receive the gold standard treatment for chronic neck pain including mobilization and modalities. In addition to the gold standard treatment the participants will receive specific stretching protocol based on their interventional group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator and outcome assessor are not aware of which treatment group the participant/patient is placed in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Control Group - Static Stretching) (Active Comparator): (Control Group - Static Stretching + Standard Treatment)
  Interventions: Other: Group A (Control Group - Static Stretching + Standard Treatment)
- Group B (Autogenic Inhibition MET) (Experimental): (Autogenic Inhibition - PIR + Standard treatment)
  Interventions: Other: Group B (Autogenic Inhibition - PIR + Standard treatment)
- Group C (Reciprocal Inhibition MET) (Experimental): (Reciprocal Inhibition - RI + Standard treatment)
  Interventions: Other: Group C (Reciprocal Inhibition - RI + Standard treatment)

INTERVENTIONS:
Other: Group A (Control Group - Static Stretching + Standard Treatment) — o Conventional Gold Standard treatment (Manual Therapy + Modalities) Conventional Static Stretching 15-30 seconds hold 3-5 repetitions (Page P, 2012) for Ant/Middle/Posterior Scaleni, Sternocleidomastoid, Levator Scapulae and Upper Trapezius Muscles.
  Arms: Group A (Control Group - Static Stretching)
Other: Group B (Autogenic Inhibition - PIR + Standard treatment) — o Conventional Gold Standard treatment (Manual Therapy + Modalities) Post Isometric Relaxation MET (3-5 reps) for Ant/Middle/Posterior Scaleni, Sternocleidomastoid, Levator Scapulae and Upper Trapezius Muscles. (Chaitow L, 2006)
  Arms: Group B (Autogenic Inhibition MET)
Other: Group C (Reciprocal Inhibition - RI + Standard treatment) — o Conventional Gold Standard treatment (Manual Therapy + Modalities) Reciprocal Inhibition MET (3-5 reps) for Ant/Middle/Posterior Scaleni, Sternocleidomastoid,Levator Scapulae and Upper Trapezius Muscles (Chaitow L, 2006)
  Arms: Group C (Reciprocal Inhibition MET)

SUMMARY:
Neck pain is among the most common musculoskeletal disorders worldwide and is an important public health issue in terms of personal wellbeing. Prevalence of neck pain show excessive variations, with a point prevalence varying between 6% and 22%, and one year prevalence ranging between 1.5-75%. Neck pain like all other mechanical disorders leads to pain, disability and decreased range of motion (ROM). Stretching is a very common exercise performed by sportsmen, elderly, in physical therapy and rehabilitation patients, thus practiced in all sorts of fitness programs. The major types of stretching included in the literature are static, dynamic and pre-contraction stretching; of which static stretching is the conventional type of stretching. The different types of pre-contraction stretching include Proprioceptive Neuromuscular Facilitation (PNF) stretching, Post Isometric Relaxation (PIR), Post Facilitation stretch (PFS) and Active Isolated Stretch (AIS). Pre-contraction stretching is also considered a part of Muscle Energy Technique (MET). Recently MET and pre-contraction stretching have been shown to have significant superiority over conventional stretching in management of mechanical neck pain, but the evidence is currently lacking regarding which of the two pre-contraction stretching protocols, namely autogenic and reciprocal inhibition is more effective than the other. A RCT will be conducted in order to find and compare the effectiveness of conventional stretching and pre-contraction stretching (autogenic inhibition and reciprocal inhibition). One Control group (conventional group) and two Experimental groups (Experimental Group A - Autogenic Inhibition & Experimental Group B - Reciprocal Inhibition) will be formed. The participants will be recruited in the study if they meet the inclusion criteria using consecutive sampling from Fauji Foundation Hospital and randomized into the three respective groups. All the groups will receive the gold standard treatment for chronic neck pain including mobilization and modalities. In addition to the gold standard treatment the participants will receive specific stretching protocol based on their interventional group

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years;
2. Neck pain on NPRS 4 to 8 (moderate cases);
3. Subacute or chronic cases (4 to 12 weeks).
4. Decreased or painful Cervical range of motion (CROM)

Exclusion Criteria:

1. Signs of serious pathology (e.g., malignancy, inflammatory disorder, infection);
2. History of cervical spine surgery in previous 12 months;
3. History of trauma or fractures in cervical spine;
4. Signs of cervical radiculopathy or myelopathy; and
5. Vascular syndromes such as VBI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Pain (Numeric Pain Rating Scale) - Change is being assessed | Pre-treatment (First day before treatment), Immediate Follow Up (After 1st treatment session) & Follow Up (After 5 days of Treatment)
  To measure the pre and post patient's perception of pain
Cervical Range of Motion (CROM) - Change is being assessed | Pre-treatment (First day before treatment), Immediate Follow Up (After 1st treatment session) & Follow Up (After 5 days of Treatment)
  To measure patient's improvement in cervical range of motion
Neck Disability Index (NDI) - Change is being assessed | Pre-treatment (First day before treatment), Immediate Follow Up (After 1st treatment session) & Follow Up (After 5 days of Treatment)
  to measure patient's pre and post functional disability
Cervical Isometric Muscle Strength (Modified Sphygmomanometer dynamometry) - Change is being assessed | Pre-treatment (First day before treatment), Immediate Follow Up (After 1st treatment session) & Follow Up (After 5 days of Treatment)
  To measure patient's improvement in Isometric Muscle Strength

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, DPT, MS-OMPT, CHPE, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Institute of Rehabilitation Sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No